CLINICAL TRIAL: NCT02385149
Title: Improving Resilience With Whole Grain Wheat
Acronym: Graandioos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: TNO (Other); Cereal Partners Worldwide (Industry); Nederlands Bakkerij Centrum (Other); Goodmills (Unknown); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL51389.081.14
Record Dates: First submitted 2015-02-19; First posted 2015-03-11 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-03

CONDITIONS: Healthy; Metabolism
Keywords: resilience; challenge test; whole grain wheat; metabolic flexibility; cardio-metabolic; liver and adipose tissue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- whole grain wheat (Experimental): 98g whole grain wheat per day for 12 weeks
  Interventions: Other: whole grain wheat
- refined wheat (Experimental): coloured refined wheat control intervention
  Interventions: Other: refined wheat

INTERVENTIONS:
Other: whole grain wheat — A twelve week intervention of 98g whole grain wheat in the form of 4 slices of bread (is in total 100g bread) and 2 servings of ready to eat cereals (RTEC, is in total 33.4g RTEC).
  Arms: whole grain wheat
Other: refined wheat — A twelve week control intervention of refined wheat in the form of 4 slices of bread (is in total 100g bread) and 2 servings of ready to eat cereals (RTEC, is in total 33.4g RTEC).
  Arms: refined wheat

SUMMARY:
This study investigates the health benefits of whole grain wheat on cardiovascular/ cardio-metabolic health, including glucose metabolism, by means of applying a mixed meal challenge. This study also investigates the health benefits of whole grain wheat (WGW) on liver- and adipose tissue health and evaluates the potential of do-it-yourself (DIY) devices in quantifying health effects in a nutritional intervention study.

DETAILED DESCRIPTION:
The study is a randomized controlled, double blind, parallel trial. A 4-week run-in period with refined wheat (RW) products will be included prior to the intervention for all subjects. Thereafter, two different treatments will be evaluated e.g. a 12-week intervention with whole grain wheat (WGW) products (98g of WGW per day) and a 12-week control intervention with RW products. Two experimental visits will be planned before and two experimental visits will be planned after the 12-week intervention period. In the first experimental visit the investigators will determine liver fat and abdominal fat distribution by magnetic resonance spectroscopy (MRS) and magnetic resonance imaging (MRI). In the second experimental visit the investigators will comprehensively phenotype the participants which will include the response to a mixed meal challenge test.

ELIGIBILITY:
The inclusion of subjects with mildly impaired cardio-metabolic risk profiles enables detection of improvements in health after WGW consumption. The investigators therefore aim to include 50 middle aged and overweight males or postmenopausal females (45-70yrs and BMI between 25-35 kg/m2) that have mildly elevated levels of cholesterol (cholesterol levels > 5 mmol/L). In case the inclusion of subjects with mildly elevated levels of total cholesterol is too difficult, normal levels of total cholesterol (< 5 mmol/L) can be accepted, but with a minimum total cholesterol level of 4.5 mmol/L.

Inclusion Criteria:

* Males or postmenopausal females (target 50: 50 for both genders) For females: menstrual cycle absent for more than 1 year
* Age 45-70yrs
* BMI between 25 and 35 kg/m2
* Signed informed consent
* Normal food habit of bread and cereal consumption

Exclusion Criteria:

* Not having a general practitioner
* Having a history of medical or surgical events that may significantly affect the study outcome
* Smoker
* Use of cholesterol lowering medication
* Mental status that is incompatible with the proper conduct of the study
* Aversion, intolerance to gluten, whole wheat or other items in the intervention products
* Alcohol consumption of > 21 glasses a week
* Abuse of drugs
* Recent use of antibiotics (<1 month prior to day 01 of the study)
* Reported weight loss or weight gain of > 5 kg in the month prior to pre-study screening
* Reported slimming or medically prescribed diet
* Reported vegan or macrobiotic life-style
* Not willing to give up blood donation during the study
* Personnel of Wageningen University, department of Human Nutrition, their partner and their first and second degree relatives
* Current participation in other research (with the exception of NQplus)
* Contraindication for MRI
* Having blood vessels that are too difficult for inserting a cannula

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in cardio-metabolic health parameters (composite) | Baseline and after 12 week intervention (at 0 and 12 weeks) , during fasting and in response to a mixed meal challenge test (at 30,60,120,240 min postprandial)
  parameters include change in cholesterol, TAG, glucose, insulin, FMD (Fasting only), pulse wave analysis (Fasting and 120, 240min postprandial), blood pressure(Fasting and 120, 240min postprandial), blood cell activation (Fasting only) and plasma markers of cardio-vascular health

SECONDARY OUTCOMES:
Change in liver-and adipose tissue health parameters (composite) | Baseline and after 12 week intervention (at 0 and 12 weeks), during fasting and in response to a mixed meal challenge test (at 30,60,120,240 min postprandial)
  parameters include change in intrahepatic lipid accumulation (by MRS, at -1 and 11 weeks), abdominal body fat distribution (by MRI, at -1 and 11 weeks), adipose tissue gene expression (adipose tissue biopsy, fasting only), blood markers of liver health
Change in do-it-yourself measure outcomes (composite) | At baseline and every two weeks during the intervention (at 0,2,4,6,8,10,12 weeks)
  DIY tests are optional and include glucose, cholesterol, blood pressure and a OGTT (only week 8). These tests are performed by the subjects.
Change in health and mood questionaire outcomes | At baseline and every two weeks during the intervention (at 0,2,4,6,8,10,12 weeks)
  health and mood questionaires (some questionaires are every 4weeks)
Change in blood markers of whole grain intake | before and after 12 week intervention (at 0 and 12 weeks)
  such as alkylresorinol

OTHER OUTCOMES:
Change in peripheral blood mononuclear cells | Baseline and after 12 week intervention (at 0 and 12 weeks), during fasting and in response to a mixed meal challenge test (at 60 and 240 min postprandial)
  gene expression
Change in markers of satiety (composite) | Baseline and after 12 week intervention (at 0 and 12 weeks, during fasting and in response to a mixed meal challenge test (at 10,30,60,120,240 min postprandial)
  parameters include questionaires and blood markers of satiety
Urine and faecal collection | Baseline and after 12 week intervention (at 0 and 12 weeks)
  To determine markers of compliance and microbiota profiling

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Afman, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen Universiteit Division of Human Nutrition, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Gijbels A, Schutte S, Esser D, Wopereis S, Gonzales GB, Afman LA. Effects of a 12-week whole-grain or refined wheat intervention on plasma acylcarnitines, bile acids and signaling lipids, and association with liver fat: A post-hoc metabolomics study of a randomized controlled trial. Front Nutr. 2022 Oct 13;9:1026213. doi: 10.3389/fnut.2022.1026213. eCollection 2022. PMID 36330140
- [Derived] van Trijp MPH, Schutte S, Esser D, Wopereis S, Hoevenaars FPM, Hooiveld GJEJ, Afman LA. Minor Changes in the Composition and Function of the Gut Microbiota During a 12-Week Whole Grain Wheat or Refined Wheat Intervention Correlate with Liver Fat in Overweight and Obese Adults. J Nutr. 2021 Mar 11;151(3):491-502. doi: 10.1093/jn/nxaa312. PMID 33188417
- [Derived] Hoevenaars FPM, Esser D, Schutte S, Priebe MG, Vonk RJ, van den Brink WJ, van der Kamp JW, Stroeve JHM, Afman LA, Wopereis S. Whole Grain Wheat Consumption Affects Postprandial Inflammatory Response in a Randomized Controlled Trial in Overweight and Obese Adults with Mild Hypercholesterolemia in the Graandioos Study. J Nutr. 2019 Dec 1;149(12):2133-2144. doi: 10.1093/jn/nxz177. PMID 31504709
- [Derived] Schutte S, Esser D, Hoevenaars FPM, Hooiveld GJEJ, Priebe MG, Vonk RJ, Wopereis S, Afman LA. A 12-wk whole-grain wheat intervention protects against hepatic fat: the Graandioos study, a randomized trial in overweight subjects. Am J Clin Nutr. 2018 Dec 1;108(6):1264-1274. doi: 10.1093/ajcn/nqy204. PMID 30541093